CLINICAL TRIAL: NCT01236092
Title: Clinical Study Comparing Traditional Physical Therapy and Alternate Therapy in Patients With Lumbar Radiculitis and Radiculopathy Secondary to Neural Compression.
Brief Title: Low Back Study to Compare Traditional Physical Therapy With Combined Therapy Protocol
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate patient enrollment
Sponsor: Michael Wilson & Associates Health Care Consulting, LLC (Industry)
Collaborators: Pneumex Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mwilson consulting, llc
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2012-07

CONDITIONS: Radiculopathy; Low Back Pain
Keywords: resolution of low back pain; show measurable improvement in disc measurement; conservative therapy vs. surgery in resolving low back pain
MeSH Terms: conditions — Radiculopathy; Low Back Pain | interventions — Vibration; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: conservative therapy - traction, vibration, exercise — 10 weeks of therapy. 3 treatments per week the first 4 weeks and 2 treatments the final 6 weeks.

SUMMARY:
The most common chronic low back pain conditions are a consequence of disc disease as well as muscular and bony etiologies. The discs degenerate and weaken, bulge and are pushed into the space containing the spinal cord or a nerve root resulting in severe pain. A common treatment is then surgery. Whole-body vibration combined with un-weighting traction and specific manual mobilization plus active therapeutic exercise seems to treat chronic low back pain by non-invasively firing muscles of the lumbar spine. The investigators are seeking to show such therapy reduces the need for surgery and significantly out performs traditional physical as the preferred conservative treatment.

DETAILED DESCRIPTION:
Patients will be placed randomly in the control group and will receive 10 weeks of standard physical therapy or in the study group and receive an equivalent 10 weeks therapy utilizing vibration, unweighting, therapeutic exercise and manual mobilization. The study uses a baseline MRI and x-rays which have shown the justification for surgical intervention and during the course of the protocol will have repeat MRI's and x-rays to determine any statistical change in the lumbar spine resulting in reduction or elimination of pain, improved range of motion, improvements in performance and reduction or elimination for the need for surgical intervention. Anatomical measures will be done comparing pre-treatment versus post-treatment and will include foraminal dimensions,disc height, canal stenosis, lumbosacral angle and facet spacing. Questionnaires will be completed during the course of the treatment and post-treatment at 6 months and one year. The final follow up phone call to the patient will be made following 24 months post initial treatment to determine the current patient status pertaining to low back pain, subsequent treatment, surgery, etc. Final study documentation will occur at that time. Intermediate results at one year will compare the control group vs. the study group for overall result differences.

ELIGIBILITY:
Inclusion Criteria:

* MRI of the lumbar spine showing symptoms and severity to qualify for surgery
* 25 to 65 years of age
* Diagnosis of low back pain for 3-12 months
* Potential surgical candidates but not mandatory

Exclusion Criteria:

* any medical or physical conditions deemed unacceptable by the participants physician or health care provider
* Evidence of progressive or debilitative medical conditions i.e. metastatic cancer, major stroke, crippling arthritis, unstable angina, orthostatic hypotension, hemiplegia, multiple sclerosis or Parkinson's disease.
* Any condition that would preclude the additional burden of a repeat MRI or preclude active involvement in the protocol or physical therapy
* Active use of tobacco products
* Prior back surgery
* Pregnancy

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Radiographic changes in the low back | 6 months following enrollment
  Anatomical measures will be done comparing pre-treatment versus post-treatment and will include foraminal dimensions, disc height, canal stenosis, lumbrosacral angle, and facet spacing.

SECONDARY OUTCOMES:
determine the percentage of patients who do not obtain relief of symptoms from either therapy and move on to surgery and determine the statistical difference between therapies. | one year following initiation of therapy
  The comparison of convervative therapies, the control group with standard physical therapy and the study group, serve as the comparitive for the success as measured by the number from each group which move to surgery within the one year.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Martz, m.d., Principal Investigator — Inland Neurosurgery and Spine
Locations (1):
- St. Luke's Rhabilitation Institute and Revita Back, Spokane, Washington, United States